CLINICAL TRIAL: NCT05730257
Title: Open-label Randomized Clinical Trial Investigating Whether Robot-Assisted Kidney Transplantation Can Reduce Surgical Complications Compared to Open Kidney Transplantation; The ORAKTx Trial
Brief Title: Study Investigating Whether Robot-assisted Surgery Can Reduce Surgical Complications Following Kidney Transplantation
Acronym: ORAKTx
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Milla Ortved, MD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-22065569; P-2022-834 (Other: Danish Data Protection Agency)
Record Dates: First submitted 2023-02-07; First posted 2023-02-15 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-10

CONDITIONS: End Stage Renal Disease; Kidney Transplant; Complications
Keywords: Kidney Transplantation; Robotic Surgery
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robot-assisted Kidney Transplantation (RAKT) (Experimental): Participants will undergo standard work-up prior to transplantation according to the KDIGO guidelines, in addition, participation in the study will require a non-contrast CT of the abdomen to exclude severe calcification of the iliac vessels.
  Participants will be managed according to the standard protocol for renal transplantation at Rigshospitalet and will follow standard pre-, peri- and post-operative care aside from operating modality. The anaestethic protocol will be tailored to suit robot-assisted surgery
  Interventions: Procedure: Robot-Assisted Kidney Transplantation
- Open Kidney Transplantation (OKT) (Active Comparator): Participants will undergo standard work-up prior to transplantation according to the KDIGO guidelines, in addition, participation in the study will require a non-contrast CT of the abdomen to exclude severe calcification of the iliac vessels.
  Participants will be managed according to the standard protocol for anaesthesia and renal transplantation at Rigshospitalet and will follow standard pre-, peri- and post-operative care aside from operating modality.
  Interventions: Procedure: Open Kidney Transplantation

INTERVENTIONS:
Procedure: Robot-Assisted Kidney Transplantation — Robot-Assisted Kidney Transplantation takes place with the patient under general anaesthesia. Several ports are placed in the lower abdomen, for the entry of the camera, surgical instruments and manuel access. The DaVinci robot is placed between the patient's legs and docked to the ports. The iliac vascular bed is prepared and a peritoneal cavity created laterally. The kidney is introduced through the handport, regional hypothermia obtained via iceslush in the cavity and the vessel lumens flushed with heparin. The vessels are blocked during suturing with the kidney graft vessels anastomosed end-to-side to the external iliac vessels. The kidney graft is placed in the retroperitoneal cavity and a ureterovesical anastomosis performed ad modem Woodruff over double J stent. The ureter is placed extra peritoneally, fascia closed in layers and the skin using intracutaneous suturing. Perioperative prophylactics entail piperacillin/tazobactam and an indwelling bladder catheter is placed.
  Arms: Robot-assisted Kidney Transplantation (RAKT)
Procedure: Open Kidney Transplantation — Open Kidney Transplantation takes place with the patient under general anaesthesia. A jockey-stick (Gibson) incision is made in the left or right iliac fossa and the peritoneum is displaced. With the kidney under hypothermia, the iliac vascular bed is prepared, the vessel lumens flushed with heparin and a vascular clamp instrument is used to block the vessels during suturing. The kidney graft vessels are anastomosed end-to-side to the external iliac vessels and the ureterovesical anastomosis performed ad modem Woodruff over a double J stent. The kidney graft is placed in the cavity and the fascia is closed in layers and the skin using intracutaneous suturing. Perioperative prophylactics entail piperacillin/tazobactam and an indwelling bladder catheter is placed.
  Arms: Open Kidney Transplantation (OKT)

SUMMARY:
The purpose of this study is to explore whether robot-assisted surgery can reduce 30-day surgical complications compared to open surgery in kidney transplantation.

Participants are adult recipients of kidney transplantation. Upon entry into the trial participants will be randomly assigned eiher open kidney transplantation or robot-assisted kidney transplantation. The participants in both groups will be treated in accordance with up-to-date guidelines and care.

Our hypothesis is that robot-assisted surgery can reduce vascular complications by 15% and/or major surgical complicatons by 20% within 30 days of kidney transplantation compared to open surgery.

DETAILED DESCRIPTION:
Kidney transplantation is the ultimate surgical treatment for end stage renal disease, and while medical transplantation therapy has developed tremendously and now allows for transplantation and long-term survival, even in seemingly incompatible donors and recipients, kidney graft survival still, to a large extent, depends on a smooth and complication-free surgical procedure. In the past decade surgical techniques have been expanded by the introduction of surgical robots to improve minimally invasive surgery and optimize post-surgical care. Previous studies suggest that robot-assisted surgery has the potential to reduce complications such as surgical site infection and blood-loss, facilitate fast-track or even ambulatory surgery for complicated procedures and recent studies suggest this may be the case for kidney transplantation too.

The aim of this trial is therefore to explore if robot-assisted surgery can reduce surgical complications following kidney transplantation compared to open surgery (standard of care) and investigate the patient trajectory following the two procedures in terms of late complications, graft function and mortality. The study design is a superiority, open-label randomized clinical trial to be conducted at Rigshospitalet, the largest transplantation centre in Denmark.

The primary outcomes consist of 1) reduction in vascular complications (graft arterial stenosis, bleeding requiring reoperation, symptomatic haematomas, renal vascular thrombosis). The rate of vascular complications is currently 17.3%. With a power set at 80% and a significance level set at 5% we hypothesize that Robot-Assisted Kidney Transplantation (RAKT) can reduce vascular complications by 15% within 30 days after transplantation compared to Open Kidney Transplantation (OKT). 2) Reduction in surgical complications Clavien-Dindo > grade 2. The rate of Clavien-Dindo >2 is currently 22.8%.

With a power set at 80% and a significance level set at 5%, we hypothesize that RAKT can reduce Clavien-Dindo >2 by 20% within 30 days after transplantation compared to OKT.

The study will randomize 106 participants with an anticipated drop-out of 10% (n=96). Immediate follow-up will be 30-days after kidney transplantation to observe occurrence of primary endpoints assessed by chart review including both in- and out-patient information. Follow-up through chart review will persist for 2 years in order to monitor long-term complications and assess secondary outcomes. Participants will be randomized with a 1:1 allocation ratio using the randomization module in REDCap with differing block sizes. Dropouts will be replaced by the same randomization number to ensure equal distribution.

The study is analysed as intention-to-treat. The primary endpoints are expected to be evaluated as percent of patients with complications compared between the two groups. Secondary outcomes will be represented descriptively and analysed according to the datatype. An interim analysis will be performed when 50% of the patients are enrolled in the study. Statistical analysis will be undertaken using R version 3.2 or later if available.

While robot-assisted kidney transplantation is still in its experimental phase, robot-assisted surgery is not and many urological procedures use robotic assistance with excellent results. With no randomized clinical trials to date comparing RAKT to OKT, this study aims to contribute with valuable evidence on the possible benefits of RAKT for both surgical outcomes and the post-operative and long-term patient trajectory.

ELIGIBILITY:
Inclusion Criteria:

* Adult recipients for renal transplantation
* Both patients in dialysis as well as pre-emptive
* For recipients of kidney grafts from deceased donors, inclusion depends on the availabilty of the robotic platform and dedicated surgical team

Exclusion Criteria:

* High degree of calcification of the iliac vessels on the level of external iliac artery defined as occurrence of longitudinal plaques on non-contrast CT-scan or other relevant radiological imaging in recipient prior to transplantation
* Highly complex vascular anatomy in the donor kidney requiring multiple anastomoses as evaluated by surgeon
* Previous kidney transplantation with later allograft nephrectomy as evaluated by the surgeon preoperatively
* Patients whose abdominal anatomy may prohibit access to and placement of graft in the iliac fossa as evaluated by the surgeon preoperatively (i.e. previous laparotomy, rectal surgery, herniotomy, current multiple kidney cysts)
* Simultaneous multiple organ transplant
* Severe comorbidities contraindicating robot-assisted surgery
* Patients who are unable to understand relevant medical information and the implications of treatment alternatives and to make an independent, voluntary decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2023-05-08 (Actual); Primary Completion 2025-10-26 (Actual); Study Completion 2027-10-26 (Estimated)

PRIMARY OUTCOMES:
Vascular complications | 30 days after surgery
  Composite outcome consisting of a) bleeding requiring reoperation, b) renal/graft vascular thrombosis, c) symptomatic hematomas d) renal/graft arterial stenosis
Surgical complications Clavien-Dindo >grade 2 | 30 days after surgery
  All postoperative complications will be recorded and graded according to the Clavien-Dindo classification with major complications defined as >grade 2.

SECONDARY OUTCOMES:
Length of Stay (LOS) | 12 months
  Duration (days) of primary hospitalization. From the date of admission until the date of discharge from hospital
Days Alive and Out of Hospital (DAOH) | 30 days after surgery
  Number of days alive and out of hospital within 30 days from surgery
Days Alive and Out of Hospital (DAOH) | 90 days after surgery
  Number of days alive and out of hospital within 90 days from surgery
Quality of Life (QOL): SF-36 | 30 days after surgery
  Patient reported health related QOL using the Short Form 36-item Health Survey
Quality of Life (QOL): SF-36 | 90 days after surgery
  Patient reported health related QOL using the Short Form 36-item Health Survey
Use of analgesics | 12 months
  Average administered dose of any opiod agent (MME/day) post surgery, during in-hospital stay
Transfusion rate | 30 days after surgery
  Total amount of red blood cells administered (units)
Kidney Function | 30 days after surgery
  30-day creatinine and estimated Glomerular Filtration Rate (eGFR). Creatinine: μmol/L. eGFR calculated according to the CKD-EPI equation
Kidney Function | 90 days after surgery
  90-day creatinine and estimated Glomerular Filtration Rate (eGFR). Creatinine: μmol/L. eGFR calculated according to the CKD-EPI equation
Kidney Function | 12 months after surgery
  1-year creatinine and estimated Glomerular Filtration Rate (eGFR). Creatinine: μmol/L. eGFR calculated according to the CKD-EPI equation
Kidney Function | 24 months after surgery
  2-year creatinine and estimated Glomerular Filtration Rate (eGFR). Creatinine: μmol/L. eGFR calculated according to the CKD-EPI equation
Delayed Graft Function (DGF) | 7 days after surgery
  Need for dialysis in the first post-operative week beyond day 0, due to lack of increase in kidney function and where the cause is not urological/surgical complications or hyperkalaemia alone
Graft loss | 30 days after surgery
  Start of permanent dialysis and/or allograft nephrectomy
Graft loss | 90 days after surgery
  Start of permanent dialysis and/or allograft nephrectomy
Graft loss | 24 months after surgery
  Start of permanent dialysis and/or allograft nephrectomy
30-day Mortality | 30 days after surgery
  30-day all cause mortality rate and cause of death
90-day Mortality | 90 days after surgery
  90-day mortality rate and cause of death
1-year Mortality | 12 months after surgery
  1-year mortality rate and cause of death
2-year Mortality | 24 months after surgery
  2-year mortality rate and cause of death
Specific urological surgical complications | 30 days after surgery
  Ureteral strictures, urinary leak, hydronephrosis, symptomatic lymphocele; including, when needed, designated intervention (nephrostomy, JJ stent, reimplantation, drain, surgery)
Late & specific urological surgical complications | 90 days after surgery
  Ureteral strictures, urinary leak, hydronephrosis, symptomatic lymphocele; including, when needed, designated intervention (nephrostomy, JJ stent, reimplantation, drain, surgery)
Late & specific urological surgical complications | 24 months after surgery
  Ureteral strictures, urinary leak, hydronephrosis, symptomatic lymphocele; including, when needed, designated intervention (nephrostomy, JJ stent, reimplantation, drain, surgery)
Time to return to work | 90 days after surgery
  Whether participants have resumed a paying job 90 days after surgery. If yes: time in months from operation until any degree of work is resumed
Recurrent urinary tract infection (UTI) | 90 days after surgery
  Culture confirmed recurrent UTI as defined by EAU guidelines (3 per year or 2 within 6 months)
Recurrent urinary tract infection (UTI) | 24 months after surgery
  Culture confirmed recurrent UTI as defined by EAU guidelines (3 per year or 2 within 6 months)
Rejection | 12 months after surgery
  Rejection within 12 months of surgery. If rejection has occurred, diagnostic category according to Banff Classification of Renal Allograft Pathology.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Roeder, MD, PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (2):
- Denmark (2):
  - Urological Research Unit, Rigshospitalet, Copenhagen, N
  - Department of Nephrology, Rigshospitalet, Copenhagen, Ø

IPD SHARING:
Plan to Share IPD: No
All study data including study protocol, statistical analysis plan, informed consent form, and clinical study report can be shared when a proper agreement is formed according to the European Union (EU) General Data Protection Regulation (GDPR) protection statement.

REFERENCES:
- [Derived] Ortved M, Dagnaes-Hansen J, Stroomberg HV, Kistorp T, Rohrsted M, Sorensen SS, Roder A. Open-label randomised clinical trial investigating whether robot-assisted kidney transplantation can reduce surgical complications compared to open kidney transplantation (ORAKTx): study protocol for a randomised clinical trial. Trials. 2025 Jan 6;26(1):8. doi: 10.1186/s13063-024-08706-5. PMID 39762978